CLINICAL TRIAL: NCT02556580
Title: Volume Kinetics for 20% Albumin in Conscious and Anesthetized Humans With and Without Inflammation
Brief Title: Volume Kinetics for 20% Albumin in Different Clinical Situations
Acronym: Albumin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sodertalje Hospital (Other)
Collaborators: University Hospital, Linkoeping (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Robert Hahn, Research Dircetor, Sodertalje Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Albumin April 2015
Record Dates: First submitted 2015-05-24; First posted 2015-09-22 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Unconscious; Inflammation
Keywords: albumin; surgery; inflammation; volume kinetics
MeSH Terms: conditions — Unconsciousness; Inflammation | interventions — galactosamine-conjugated serum albumin-conjugated-(rhodamine X)20; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conscious healthy volunteers (Active Comparator): Intervention: intravenious infusion Drug: albumin 20%
  Interventions: Drug: Albumin 20%
- Surgery under general anesthesia (Experimental): Intervention: intravenious infusion Drug: albumin 20%
  Interventions: Drug: Albumin 20%
- Post-surgical inflammation (Experimental): Intervention: intravenious infusion Drug: albumin 20%
  Interventions: Drug: Albumin 20%

INTERVENTIONS:
Drug: Albumin 20% — Intervention: intravenious infusion Drug: albumin
  Other Names: Albumin in healthy volunteers

SUMMARY:
The study aims to determine the degree of plasma volume expansion and the half-life of the plasma volume expansion when 3 mL/kg of hyperoncotic (20%) albumin if infused over 30 minutes in conscious healthy volunteers, in patients undergoing surgery under general anesthesia, and on the day after major surgery when the patient is in a post surgical inflammatory state. The study also examines the increase in the plasma colloid osmotic pressure as a result of this infusion and its possible influence on markers of kidney damage.

DETAILED DESCRIPTION:
15 volunteers, 15 patients undergoing surgery and 15 patients in the post-surgical phase will be recruited for this study because they have different degrees of vasodilatation and inflammation, which are factors of potential importance to the effectiveness of plasma volume expansion with albumin 20%. Hyperoncotic albumin should logically recruit fluid from the interstitial fluid space, but this possibility has recently been questioned in the "revised Starling equation".

The degree of plasma volume expansion and also the half-life will be estimated by population volume kinetics which uses serial analyses of the blood hemoglobin concentration and a summary measure of the excreted urine during the 5-hour experiment to calculate these outcome measures.

There is a risk that hyperoncotic solutions cause pre-renal anuria due to the rise in plasma oncotic pressure. As a safety measure we will assess the plasma oncotic pressure and relevant biomarkers of renal function during the experiments. The experiments will be ended with a slow infusion of 1 L of Ringer´s acetate to dilute any raised oncotic pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Patients in ASA classes I-II scheduled for surgery.

Exclusion Criteria:

* Expected major hemorrhage during surgery.
* Blood hemoglobin concentration of < 10 g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Degree of plasma volume expansion | 5 hours
  Calculated by volume kinetics

SECONDARY OUTCOMES:
Increase in plasma oncotic pressure | 5 hours
  Measured by oncometer
Possible effect on biomarkers of kidney injury | 5 hours
  Urinary albumin excretion (unit: mmol of albumin per mmol of urinary creatinine) and urinary neutrophil gelatinase-associated lipocalin (NGAL) excretion (unit: µg/L per mmol of creatinine).
Half-life of plasma volume expansion | 5 hours
  Calculated from the restoration of the diluted blood hemoglobnin concentration

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Hahn, MD, PhD, Principal Investigator — Research Director, Södertälje sjukhus
Locations (2):
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data from the volunteer and postoperative patients are available in March 2018. The intraoperative patients are still being recruited
Access Criteria: Contact the Project Leader

REFERENCES:
- [Background] Hedin A, Hahn RG. Volume expansion and plasma protein clearance during intravenous infusion of 5% albumin and autologous plasma. Clin Sci (Lond). 2005 Mar;108(3):217-24. doi: 10.1042/CS20040303. PMID 15538944
- [Background] Woodcock TM, Woodcock TE. Revised Starling equation predicts pulmonary edema formation during fluid loading in the critically ill with presumed hypovolemia. Crit Care Med. 2012 Sep;40(9):2741-2; author reply 2742. doi: 10.1097/CCM.0b013e31825ae6c9. No abstract available. PMID 22903119
- [Background] Wiedermann CJ, Dunzendorfer S, Gaioni LU, Zaraca F, Joannidis M. Hyperoncotic colloids and acute kidney injury: a meta-analysis of randomized trials. Crit Care. 2010;14(5):R191. doi: 10.1186/cc9308. Epub 2010 Oct 28. PMID 21029460
- [Derived] Gunnstrom M, Zdolsek JH, Hahn RG. Plasma Volume Expansion and Fluid Kinetics of 20% Albumin During General Anesthesia and Surgery Lasting for More Than 5 Hours. Anesth Analg. 2022 Jun 1;134(6):1270-1279. doi: 10.1213/ANE.0000000000005802. Epub 2021 Nov 18. PMID 34797221